CLINICAL TRIAL: NCT01605526
Title: A Multi-center, Open-label Phase IB Study of Escalating Doses of RO5045337, an Oral Small Molecule MDM2 Antagonist, in Combination With Doxorubicin in Patients With Soft Tissue Sarcoma
Brief Title: A Study of RO5045337 in Combination With Doxorubicin in Patients With Soft Tissue Sarcoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP28021; 2011-006279-21 (EudraCT Number)
Record Dates: First submitted 2012-05-04; First posted 2012-05-25 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Doxorubicin

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: RO5045337; Drug: doxorubicin

INTERVENTIONS:
Drug: RO5045337 — Multiple escalating oral doses, Days 1-5 (1-3) of each 28-day cycle, up to 6 cycles
Drug: doxorubicin — 60 mg/m2 (75 mg/m2, 50 mg/m2) iv on Day 1 of each 28-day cycle, up to 6 cycles

SUMMARY:
This multicenter, open-label, Phase 1b study will evaluate the safety, pharmacokinetics and efficacy of RO5045337 in combination with doxorubicin in patients with soft tissue sarcoma. Cohorts of patients will receive escalating doses of RO5045337 orally on Days 1-5 (1-3) of each 28-day cycle in combination with doxorubicin 60 mg/m2 intravenously on Day 1 of each cycle for up to 6 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Histologically or cytologically confirmed soft tissue sarcoma
* Evaluable disease according to RECIST version 1.1 criteria
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1
* Eligible for doxorubicin therapy
* Acute toxicities from prior anti-tumor therapy, surgery or radiotherapy must have resolved to NCI-CTCAE Grade </= 1 prior to start of study
* Adequate bone marrow, hepatic and renal function
* Patients with stable CNS metastases are eligible

Exclusion Criteria:

* Previous treatment with limiting doses of doxorubicin
* Patients receiving any other investigational or commercial agents or therapies administered with the intention to treat their malignancy or other ailment </= 28 days from Day 1 dosing on study treatment
* History of seizure disorders or unstable CNS metastases
* Severe and/or uncontrolled medical conditions or other conditions that could affect the participation in the study
* Pregnant or breastfeeding women
* HIV positive patients who are currently receiving combination anti-retroviral therapy
* Patients with known coagulopathy, platelet disorder or history of non-drug induced thrombocytopenia
* Patients receiving oral or parenteral anti-coagulants/anti-platelet agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose/dose-limiting toxicities | approximately 12 months
Safety: Incidence of adverse events | approximately 12 months

SECONDARY OUTCOMES:
Pharmacokinetics of RO5045337 and doxorubicin in combination therapy: Area under the concentration-time curve (AUC) | Pre-dose and up to 72 hours post-dose Days 1 and 5 of Cycle 1
Pharmacodynamics: Serum macrophage inhibitory cytokine-1 (MIC-1) levels | Pre-dose and up to 72 hours post-dose on Days 1 and 5 of Cycle 1

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (9):
- United States (5):
  - Santa Monica, California
  - Boston, Massachusetts
  - Hackensack, New Jersey
  - Philadelphia, Pennsylvania
  - Salt Lake City, Utah
- France (4):
  - Bordeaux
  - Lyon
  - Toulouse
  - Villejuif